CLINICAL TRIAL: NCT06695806
Title: Measurement and Evolution of the Intolerance to Uncertainty in Osteopaths and Osteopathic Students: a Longitudinal Study
Brief Title: Measurement of the Intolerance to Uncertainty in Osteopaths
Status: Enrolling by invitation | Type: Observational
Sponsor: Institut des Hautes Etudes Osteopathiques de Nantes (Other)
Collaborators: ad hoc lab (Unknown); CEESO paris (Unknown); IOR B (Unknown)
Responsible Party: Sponsor
Other Study IDs: MICO
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cognition of Osteopath

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- osteopath: Participants should be osteopaths or students in osteopathy. They need to understand french and give their consent before answering questionnaire.

SUMMARY:
Clinical reasoning is a challenging, complex, multi-dimensional, essentially introspective and poorly understood cognitive process, as well as a crucial skill for osteopaths and health professionals. It can be agreed that this includes diagnosing the patient's condition, making therapeutic decisions to improve that condition, and the practitioner's ability to assess the patient's prognosis. Individual clinical expertise is acquired through experience. Each healthcare professional develops their own approach to problem-solving and decision-making, influenced by factors such as personality, preferences, clinical perception, and professional practices. It is important to be aware that certain factors can influence their judgement and potentially affect the quality of their work. It is possible that certain factors may influence their judgement and potentially lead to errors in their decision-making, as they can be influenced by cognitive biases such as intolerance of uncertainty. Uncertainty intolerance is defined as a personal disposition characterised by negative beliefs about uncertainty and its consequences, coupled with an underlying apprehension about the unknown. Uncertainty affects the behaviour of individuals by creating a need for certainty, which in turn affects the clinical reasoning and decision-making of healthcare professionals.

The objective of this study is to assess the level of intolerance to uncertainty among osteopathic students and osteopaths using an online self-report questionnaire. A second questionnaire will be sent out six months after the first, allowing to assess individual changes in this intolerance over time. Furthermore, the impact of being a graduate, anxiety and the type of osteopath responding to the questionnaire will be examined. The final measure will be evaluated using a classification method called latent class analysis. This will be based on responses to questions about their relationship to evidence-based practice, dogmatism and their thoughts about the impact of osteopathic treatment.

The aim of this study is to carry out a psychometric validation of the intolerance to uncertainty questionnaire on a population of osteopaths.

ELIGIBILITY:
Inclusion Criteria:

* Student in osteopathy (3rd, 4th or 5th year) or have a diploma in osteopathy
* Provide an informed consent

Exclusion Criteria:

* Patients refusing to take part in the study.
* Pregnant women
* Patients under legal protection
* Patients who are protected adults or adults unable to express their consent.
* Withdrawal of consent to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Students are selected in three different fench schools of osteopathy, and osteopaths are selected from among former graduates of these schools.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Intolerance to uncertainty | at enrollement
  Total score of the questionnaire: Intolerance of Uncertainty Scale in Health (IUS-12-H), consisting of 12 questions. Participants answer on a Likert scale ranging from "not at all characteristic of me" (1), "somewhat characteristic of me" (2), "somewhat characteristic of me" (3), "very characteristic of me" (4), and "very characteristic of me" (5). The score ranges from 12 (no intolerance of uncertainty) to 60 (great intolerance of uncertainty).

SECONDARY OUTCOMES:
Change in Intolerance to uncertainty | From enrollement to the second assessment, six mounth later.

CONTACTS AND LOCATIONS:
Locations (1):
- IDHEO nantes, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From publication of the results to 5 years after this publication.
Access Criteria: By emailing the corresponding author with a research plan.